CLINICAL TRIAL: NCT01970215
Title: A Multi-Centre, Randomised, Double-Blind, Placebo-Controlled, Parallel-Group Study of TA-8995 in Patients With Mild Dyslipidaemia, Alone and In Combination With Statin Therapy
Brief Title: TA-8995: Its Use in Patients With Mild Dyslipidaemia (TULIP)
Acronym: TULIP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Xention Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TA-8995-03; 2012-005643-24 (EudraCT Number)
Record Dates: First submitted 2013-10-21; First posted 2013-10-28 (Estimated); Last update posted 2014-08-21 (Estimated); Status verified 2014-08

CONDITIONS: Dyslipidemia
MeSH Terms: conditions — Dyslipidemias | interventions — TA-8995; Atorvastatin; Rosuvastatin Calcium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (9):
- Group 1 (Placebo Comparator): TA-8995 0mg (placebo) & placebo statin
  Interventions: Drug: TA-8995 0mg (placebo); Drug: Placebo Statin
- Group 2 (Experimental): TA-8995 1mg & placebo statin
  Interventions: Drug: TA-8995; Drug: Placebo Statin
- Group 3 (Experimental): TA-8995 2.5mg & placebo statin
  Interventions: Drug: TA-8995; Drug: Placebo Statin
- Group 4 (Experimental): TA-8995 5mg & placebo statin
  Interventions: Drug: TA-8995; Drug: Placebo Statin
- Group 5 (Experimental): TA-8995 10mg & placebo statin
  Interventions: Drug: TA-8995; Drug: Placebo Statin
- Group 6 (Active Comparator): TA-8995 0mg (placebo) & atorvastatin 20mg
  Interventions: Drug: Atorvastatin; Drug: TA-8995 0mg (placebo)
- Group 7 (Active Comparator): TA-8995 10mg & atorvastatin 20mg
  Interventions: Drug: TA-8995; Drug: Atorvastatin
- Group 8 (Active Comparator): TA-8995 0mg (placebo) & rosuvastatin 10mg
  Interventions: Drug: Rosuvastatin; Drug: TA-8995 0mg (placebo)
- Group 9 (Active Comparator): TA-8995 10mg & rosuvastatin 10mg
  Interventions: Drug: TA-8995; Drug: Rosuvastatin

INTERVENTIONS:
Drug: TA-8995
  Arms: Group 2; Group 3; Group 4; Group 5; Group 7; Group 9
Drug: Atorvastatin
  Arms: Group 6; Group 7
Drug: Rosuvastatin
  Arms: Group 8; Group 9
Drug: TA-8995 0mg (placebo)
  Arms: Group 1; Group 6; Group 8
Drug: Placebo Statin
  Arms: Group 1; Group 2; Group 3; Group 4; Group 5

SUMMARY:
The primary objective of this study is to evaluate the efficacy of different doses of TA-8995, a cholesteryl ester transfer protein (CETP) inhibitor, on the elevation of high-density lipoprotein cholesterol (HDL-C) and reduction of low-density lipoprotein cholesterol (LDL-C), alone and in combination with statin therapy.

The secondary objectives of this study are to determine the safety and tolerability of TA-8995 in patients with mild dyslipidaemia.

ELIGIBILITY:
Inclusion Criteria:

* Fasting LDL-C levels >2.5 mmol/L and <4.5 mmol/L, HDL-C levels <1.8 mmol/L and >0.8 mmol/L, and TG levels <4.5 mmol/L after run in or washout of existing therapies
* Not on lipid-altering therapy at screening or on lipid-altering treatment regimens at screening

Exclusion Criteria:

* Body mass index >32 kg/m2;
* Participation in another clinical study involving an investigational or marketed drug within 30 days prior to enrolment (Visit 2);
* Any clinical manifestation of atherosclerotic vascular disease;
* Diagnosis of type 1 diabetes;
* Uncontrolled type 2 diabetes: haemoglobin A1c >8%;
* Uncontrolled hypertension: sitting systolic blood pressure >160 mmHg and/or sitting diastolic blood pressure >90 mmHg;
* History of hyperaldosteronism;
* Active muscle disease or persistent creatine kinase concentration >3 × the upper limit of normal (ULN). One retest will be allowed after 1 week to verify the result;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 364 (Actual)
Dates: Start 2013-08; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
The co-primary efficacy endpoints are the percentage changes in both HDL-C and LDL-C levels at Week 12 compared to baseline. | 12 weeks

CONTACTS AND LOCATIONS:
Locations (17):
- Denmark (5):
  - H:S Amager Hospital, Copenhagen
  - Sydvestjysk Sygehus, Esbjerg
  - Herlev University Hospital, Herlev
  - Hvidovre Hospital, Hvidovre
  - Regionshopitalet - Silkeborg, Silkeborg
- Netherlands (12):
  - EB FlevoResearch B.V, Almere Stad
  - Andromed Amsterdam, Amsterdam
  - Andromed Leiden, Amsterdam
  - Academic Medical Centre, Amsterdam-Zuidoost
  - Andromed Breda B.V, Breda
  - Andromed Eindhoven, Eindhoven
  - Andromed Noord B.V, Groningen
  - Andromed Zoetermeer, Leiderdorp
  - Andromed Rotterdam BV, Rotterdam
  - Albert Schweitzer Ziekenhuis, Sliedrecht
  - Andromed Oost, Velp
  - Praktijk Zwijndrecht, Zwijndrecht

REFERENCES:
- [Derived] Martin SS, Ditmarsch M, Simmons M, Alp N, Turner T, Davidson MH, Kastelein JJP. Comparison of low-density lipoprotein cholesterol equations in patients with dyslipidaemia receiving cholesterol ester transfer protein inhibition. Eur Heart J Cardiovasc Pharmacother. 2023 Feb 2;9(2):148-155. doi: 10.1093/ehjcvp/pvac056. PMID 36307922
- [Derived] van Capelleveen JC, Kastelein JJ, Zwinderman AH, van Deventer SJ, Collins HL, Adelman SJ, Round P, Ford J, Rader DJ, Hovingh GK. Effects of the cholesteryl ester transfer protein inhibitor, TA-8995, on cholesterol efflux capacity and high-density lipoprotein particle subclasses. J Clin Lipidol. 2016 Sep-Oct;10(5):1137-1144.e3. doi: 10.1016/j.jacl.2016.06.006. Epub 2016 Jun 25. PMID 27678430
- [Derived] Hovingh GK, Kastelein JJ, van Deventer SJ, Round P, Ford J, Saleheen D, Rader DJ, Brewer HB, Barter PJ. Cholesterol ester transfer protein inhibition by TA-8995 in patients with mild dyslipidaemia (TULIP): a randomised, double-blind, placebo-controlled phase 2 trial. Lancet. 2015 Aug 1;386(9992):452-60. doi: 10.1016/S0140-6736(15)60158-1. Epub 2015 Jun 2. PMID 26047975